CLINICAL TRIAL: NCT04697394
Title: To Examine Whether a Complex Intervention Protocol Decreases Toxicity in Patients Following Radiotherapy or Surgery for Colorectal Cancer. Stage 1- Feasibility of Electronic Data Collection
Brief Title: CITRuS Stage 1; Feasibility
Acronym: CITRuS1
Status: Completed | Type: Observational
Sponsor: Royal Surrey County Hospital NHS Foundation Trust (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government); The Clatterbridge Cancer Centre NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: CITRuS v3.0
Record Dates: First submitted 2021-01-05; First posted 2021-01-06 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Colorectal Cancer
Keywords: Colorectal; Cancer; PROMs; Patient Reported Outcome Measures; Electronic; Complex Intervention Protocol
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Bowel cancer is the third most common cancer occurring in the UK. Treatment usually involves surgery, often with chemotherapy or radiotherapy. In some cases radiotherapy can be used instead of surgery, especially if surgery may cause a higher risk of symptoms or a colostomy bag. Currently, the medical team collects information on patients' symptoms before and after treatment by direct questions in a clinic setting. It's recognised that patient-reported symptoms often differ from doctor-documented symptoms. This leads to inaccuracies in doctors' descriptions of the effects of cancer or treatment to patients. Patients told us an accurate description of expected symptoms is important when they are choosing their treatment.

Patient-Reported outcomes measures (PROMs) may help us identify what affects the QoL after treatment and develop ways to improve it. The primary aim of the trial is to evaluate whether patients find it acceptable to use electronic data collection to assess their symptoms. Many bowel cancer patients are elderly and they may find electronic data system collection more challenging. The secondary aim is to identify which symptoms impact QoL. This will lead to the development of treatments to manage these symptoms which will be assessed in CITRuS2.

All patients diagnosed with bowel cancer are entered into the colorectal database to determine the effectiveness of cancer treatments and outcomes. Participants will electronically answer questionnaires at study entry and during follow up. The questions are related to health and well-being with a holistic approach. The questions will take approximately 45 minutes to answer the first time and then 15 minutes thereafter. Following consent, participants gain access to their clinical details on the database. Then they can use a computer, laptop, tablet or smart phone to access a webpage and answer questions at monthly intervals over a 2 year period. Email reminders will be sent to prompt log on.

This may help discover how bowel cancer and its treatment affect patients and their lives. This may help doctors describe the effects of treatment more accurately to future patients. It may also help doctors identify which patients need extra help or support through their treatment. Electronic data may allow patterns to be identified that may not be seen by doctors until a later stage. This may enable earlier treatment resulting in less time with symptoms, which could be physically and economically beneficial.

DETAILED DESCRIPTION:
Currently, the medical team collects information on patients' symptoms before and after cancer treatment in response to direct questioning in outpatient clinics. It's recognised that patient-reported symptoms often differ from doctor-documented symptoms. Over time, this leads to inaccuracies in doctors' descriptions of the effects of cancer or its treatment to patients. Patients told us accurate description of expected symptoms is important when they are choosing which treatment to have.

This study will use an electronic database to allow colorectal cancer patients to view their treatment records. Patients will answer questions at study entry and at set intervals during treatment and follow-up. The questions are related to health and well-being. The questionnaires are patient reported outcome measures (PROMs) which have been used in paper format in trials with many patients internationally.

The information the patients give us will help doctors describe treatment effects more accurately to future patients and to identify patients who may need extra support during or after their treatment. Electronic data collection allows patterns to be identified that may not be seen by doctors until a later stage. The symptoms identified in this study will be used to develop treatments that may benefit future patients. The electronic database will be used identify the need for intervention then to deliver the recommended treatments to patients automatically when they are identified. For example, if questionnaire responses show a patient has an unplanned loss of 3% of their body weight an information sheet on increasing calorie intake and eating well with a small appetite would be emailed to them and a dietician alerted so a follow up call could be made two weeks later.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with colorectal cancer from the 5 participating centres (Guilford, Clatterbridge, Nottingham, Queens Hospital and Hull)
* No distant metastases
* Patients due to undergo surgery or radiotherapy as a definitive treatment
* ≥ 18 years of age. No maximum age.
* The ability to complete an internet based English written questionnaire either from their home or on a portable electronic device
* Patients to have read the patient information sheet and have electronically signed the informed consent
* Follow-up in clinic possible

Exclusion Criteria:

* Patient choice
* < 18 years of age
* Evidence of metastatic disease
* History of other cancer less than five years ago, excluding non-melanoma skin cancer
* Evidence of metastatic disease-patients not undergoing surgery or radiotherapy as a definitive treatment
* The inability to complete an internet based English written questionnaire at home or on a portable electronic device
* Patient with history of poor compliance or current or past psychiatric conditions that would interfere with compliance to the study protocol or cause further psychological distress.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over 18 years of age, any sex and any ethnicity who have been diagnosed with a colorectal adenocarcinoma with no evidence of distant metastases and will be receiving radiotherapy and/or surgical treatment.
Sampling Method: Probability Sample
Enrollment: 380 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2024-07-26 (Actual); Study Completion 2024-07-26 (Actual)

PRIMARY OUTCOMES:
Ability to complete the web-based electronic questionnaires online outside of the hospital setting. | 2 years
  Colorectal patients ability to electronically complete patient reported outcome measures
Continuous retention of patients completing electronic data. | 2 years
  Sustained retention of electronic data collection from colorectal patients over a 2 year period

SECONDARY OUTCOMES:
Symptom cluster identification | 1 year
  Identification of symptom clusters in the electronic data to use for part 2 of the study

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Stewart, DM, MRCP, FRCR, Principal Investigator — Consultant Clinical Oncologist, Royal Surrey County Hospital
Locations (1):
- Royal Surrey County NHS Foundation Trust, Guildford, Surrey, United Kingdom